CLINICAL TRIAL: NCT06521281
Title: The Effect of Chan-Chuang Qigong on Fatigue, Exercise Capacity and Quality of Life in Patients With Heart Failure
Brief Title: The Effect of Chan-Chuang Qigong on Fatigue, Exercise Capacity and Quality of Lifpatients With Heart Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chia-Lin Hsieh (Other)
Responsible Party: Sponsor-Investigator, Chia-Lin Hsieh, Assistant hand nurse, Cheng-Hsin General Hospital
Organization: Cheng-Hsin General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CHGH-IRB（946）111-25
Record Dates: First submitted 2024-07-10; First posted 2024-07-25 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Heart Failure NYHA Class II

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- qigong group (Experimental): Patients in qigong group was given twice daily, every 15 minutes Chan-Chuang qigong
  Interventions: Behavioral: Chan-Chuang qigong
- control group (No Intervention): control group received the regular care for heart failure patients

INTERVENTIONS:
Behavioral: Chan-Chuang qigong — Twice daily, every 15 minutes Chan-Chuang qigong
  Arms: qigong group

SUMMARY:
This study aimed to investigate the impact of Chan-Chuang Qigong on fatigue, exercise capacity, quality of life, and heart function in heart failure patients. The study recruited 72 heart failure patients from a medical center in northern Taiwan for an experimental study. The participants were randomly divided into two groups: patients in experimental group was given twice daily, every 15 minutes Chan-Chuang qigong, control group received the regular care for heart failure patients. Data was collected using the Piper Fatigue Scale, a six-minute walking test, and the Minnesota Living with Heart Failure Questionnaire before the intervention as the baseline, and at the 4th, 8th, and 12th weeks during the intervention. It is hoped that through this study, we can understand the effect of Chan-Chuang qigong on improving fatigue, exercise capacity and quality of life in patients with heart failure, and provide an additional choice and reference for the treatment and care of patients with heart failure in the future, and recommend future treatment of heart failure.

ELIGIBILITY:
Inclusion Criteria:

1. at least 20 years of age.
2. Cardiology specialist diagnoses heart failure based on clinical examination
3. Heart failure classified as New York Heart Association class II (NYHA II)
4. Left ventricular ejection volume <50% (HFmrEF and HFrEF)
5. According to the doctor's assessment, it is not appropriate to exercise
6. Clear consciousness and ability to communicate
7. Agree to participate in this study after explanation and sign the consent form

Exclusion Criteria:

1. Renal failure treated with hemodialysis
2. Severe arrhythmias, such as third-degree atrioventricular block, frequent ventricular pulses and heartbeats greater than 130 beats/min at rest
3. About to undergo coronary interventional surgery or cardiac surgery within 3 months
4. Coronary interventional surgery or cardiac surgery in the past 3 months

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2022-09-16 (Actual); Primary Completion 2023-11-25 (Actual); Study Completion 2023-11-25 (Actual)

PRIMARY OUTCOMES:
Use the Chinese version of Piper fatigue scale to assess fatigue levels. | before the intervention as the baseline, and at the 4th, 8th, and 12th weeks during the intervention
  Use the Chinese version of Piper fatigue scale.There are 16 questions in total. Based on a four-point Likert scale, the minimum score is 16 points and the maximum total score is 64 points. The higher the score, the more serious the fatigue.
Use the Six Minute Walking Distance (6MWD) to assess the patient's exercise capacity. | before the intervention as the baseline, and at the 4th, 8th, and 12th weeks during the intervention
  Use the Six Minute Walking Distance (6MWD) to assess the patient's exercise tolerance by measuring the distance the patient walks in a straight line on a surface above 30 meters for 6 minutes.
Use the Chinese version of the Minnesota Heart Failure Quality of Life to assess quality of life. | before the intervention as the baseline, and at the 4th, 8th, and 12th weeks during the intervention
  Use the Chinese version of the Minnesota Heart Failure Quality of Life Questionnaire.There are 21 questions in total, scored from 0 to 5, with a total score of 105. The higher the score, the more serious the impact of the disease on life.

SECONDARY OUTCOMES:
heart function-Left ventricular ejection volume | before the intervention as the baseline, and the twelfth week of intervention respectively
  Left ventricular ejection volume were collected by reviewing medical records.
heart function-Serum NT-pro BNP values | before the intervention as the baseline, and the twelfth week of intervention respectively
  Serum NT-pro BNP values were collected by reviewing medical records.

CONTACTS AND LOCATIONS:
Locations (1):
- Hsieh Chia Lin, Taipei, Taiwan